CLINICAL TRIAL: NCT04710927
Title: The Use of Silver Diamine Fluoride and Papain-Based Gel for Management of MIH-affected Molar in Paediatric Patients: A Randomised Controlled Trial
Brief Title: Silver Diamine Fluoride and Papain-Based Gel for Management of MIH-affected Molar in Paediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Tengku Nurfarhana Nadirah Bt Tengku Hamzah, Lecturer in Paediatric Dentistry, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF CD1912/0061/20155(P)
Record Dates: First submitted 2020-12-27; First posted 2021-01-15 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Molar Incisor Hypomineralization; Dental Caries; Hypomineralization of Enamel
Keywords: molar incisor hypomineralization; silver diamine fluoride; deproteinizing agent
MeSH Terms: conditions — Molar Hypomineralization; Dental Caries; Dental Enamel Hypomineralization

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant were not informed regarding intervention given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- High Viscosity GIC (HVGIC) (Active Comparator): Group 1
  Interventions: Device: High Viscosity Glass Ionomer Cement (HVGIC)
- Silver Diamine Fluoride (SDF) + HVGIC (Experimental): Group 2
  Interventions: Device: Silver Diamine Fluoride
- Papain based gel + SDF + HVGIC (Experimental): Group 3
  Interventions: Device: Papain-Based Gel

INTERVENTIONS:
Device: Silver Diamine Fluoride — A single application of SDF 38% (Riva Star) on dry affected molar for 1 minute and immediately restored using HVGIC
  Other Names: Riva Star
  Arms: Silver Diamine Fluoride (SDF) + HVGIC
Device: Papain-Based Gel — Papain based Gel (Papacare Duo) will be applied to the MIH affected molar for 60 seconds and repeated if required. The molar will be treated with SDF and restored using HVGIC
  Other Names: Papacare Duo
  Arms: Papain based gel + SDF + HVGIC
Device: High Viscosity Glass Ionomer Cement (HVGIC) — The molar will be restored with HVGIC
  Other Names: Riva Self Cure HV
  Arms: High Viscosity GIC (HVGIC)

SUMMARY:
Molar incisor hypomineralization (MIH) is a developmental defect of enamel affecting the first permanent molar and frequently the incisors with a prevalence of 16-16.9% in Malaysia. They presented with many problems such as hypersensitivity, increase susceptibility of caries, need for recurrent complex dental treatment, and difficulty to achieve pain control. Silver Diamine Fluoride is a new form of topical fluoride that has been extensively used and recommended for the management of caries in children and adolescents. The influence of organic material removal from artificial dentine lesions by means of surface pre-treatment with deproteinizing agent show favoring result of its use on subsequent remineralization with and without fluoride. The purpose of this trial is to study the clinical outcome of SDF and papain based gel on hypomineralized teeth restored with HVGIC.

DETAILED DESCRIPTION:
This is a three-arm parallel randomized controlled trial and will be performed in participants between the age of 5 to 15 years presented with hypomineralised molar of MIH in origin.

Clinical assessment, radiograph, and photographs will be taken for assessment. Patients that fulfilled the inclusion criteria will be invited to the study. After that, the patient will be explained and a Patient Information Sheet (PIS) will be given. Once consent obtained and the patient randomly allocated for the treatment group, treatment will be done as below:

For group 1, any caries if present will be removed using a hand instrument. The tooth then will be filled with High Viscous Glass Ionomer Cement (HVGIC) following the manufacturer's instruction. If the participant is assigned to group 2, after caries has been removed using a hand instrument, silver diamine fluoride (SDF) will be applied for 1 minute on the affected area prior to restoration with HVGIC following the manufacturer's instruction. If the participant is assigned to group 3, papain-based gel (Papacare Duo) will be applied as a deproteinizing agent, caries will be removed using a hand instrument if present. Then, silver diamine fluoride will be applied for 1 minute on the affected area prior to restoration with HVGIC following the manufacturer's instruction.

The patient will be followed up after 6 and 12 months. The teeth and restoration will be assessed clinically by an assessor that is not involved in the provision of treatment. Sign and symptom of pain, tenderness to percussion, presence of swelling or fistula, the scale of sensitivity using Schiff Cold Air Sensitivity Scale (SCASS), quality if restorative assessment using Atraumatic Restorative Treatment (ART) Index

ELIGIBILITY:
Inclusion Criteria:

1. Healthy with ability to comprehend instruction and perform oral hygiene care independently
2. Hypomineralised First Permanent Molar with:

2.1 Post Eruptive Breakdown (Code 3)

2.2 Atypical restoration (Code 4) which is unsatisfactory or with secondary caries that require replacement

2.3 Atypical caries (Code 5) with enamel breakdown

Exclusion Criteria:

1. Patient with silver allergy
2. First Permanent Molar with:

2.1 Non-MIH defect

2.2 White, creamy demarcated yellow or brown opacities (Code 2)

2.3 Good satisfactory atypical restoration (Code 4)

2.4 Atypical caries (Code 5) with pulpal involvement -Irreversible pulpitis and pulpal necrosis

2.5 Extensive coronal breakdown (Code 7)

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tengku Nurfarhana Bt Tengku Hamzah, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Dentistry, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period : 1st December 2019 to 6th October 2020 Location: Paediatric Dental Clinic, Faculty of Dentistry, University of Malaya, Kuala Lumpur, Malaysia
Pre-assignment Details: For this study, Molar Incisor Hypomineralisation (MIH) affected molar was used as unit prior assignment to intervention groups. The reason for this, data collections were affected by the peak of Coronavirus disease (COVID-19) pandemic with movement control orders enforcement for months in Malaysia. Due to this problem, one participants may had one to four molars (teeth) affected with MIH and be assigned into more than 1 intervention groups. Total participants for this study was 38 participants.
Units Other Than Participants: number of MIH affected molars
Groups:
- High Viscosity Glass Ionomer Cement (HVGIC) (Group 1): High Viscosity Glass Ionomer Cement: The MIH affected molar will be restored with HVGIC
- Silver Diamine Fluoride(SDF) + HVGIC (Group 2): Silver Diamine Fluoride(SDF): A single application of SDF 38% (Riva Star) on dry affected molar for 1 minute and immediately restored using HVGIC
- Papain Based Gel + SDF + HVGIC (Group 3): Papain-Based Gel: Papain based Gel (Papacare Duo) will be applied to the MIH affected molar for 60 seconds and repeated if required. The molar will be treated with SDF and restored using HVGIC
Period: Overall Study
Arm/Group | High Viscosity Glass Ionomer Cement (HVGIC) (Group 1) | Silver Diamine Fluoride(SDF) + HVGIC (Group 2) | Papain Based Gel + SDF + HVGIC (Group 3)
Started | 18; 21 number of MIH affected molars (Total of 10 participants in treatment arm/group 1 had more than 1 treatment interventions (6 participants had 2 treatment interventions and 4 participants with 3 treatment interventions). Only 8 participants had 1 treatment intervention. However, 3 participants from a total of 18 participants had 2 teeth assigned into treatment arm/group 1 regardless having assigned to single or more than 1 treatment group (2 and 3 treatment interventions).) | 19; 21 number of MIH affected molars (Total of 12 participants in treatment arm/group 2 had more than 1 treatment interventions (8 participants had 2 treatment interventions and 4 participants with all 3 treatment interventions). Only 7 participants had 1 treatment intervention. However, 2 out of 8 participants from 2 treatment interventions had 2 teeth assigned for treatment arm/group 2.) | 20; 21 number of MIH affected molars (Total of 11 participants in treatment arm/group 3 had more than 1 treatment interventions (7 participants had 2 treatment interventions and 4 participants with 3 treatment interventions). Only 9 participants had 1 treatment intervention. However, 1 out of 4 participants from 3 treatment interventions had 2 teeth assigned for treatment arm/group 3.)
6 Months | 15; 18 number of MIH affected molars (As units: 3 MIH affected molars failures to attend follow up at 6 months which involved 3 participants) | 16; 17 number of MIH affected molars (As units: 4 MIH affected molars failures to attend follow up at 6 months which involved 3 participants) | 16; 17 number of MIH affected molars (As units: 4 MIH affected molars failures to attend follow up at 6 months which involved 4 participants)
12 Months | 11; 13 number of MIH affected molars (As units: 8 MIH affected molars failures to attend follow up at 12 months which involved 7 participants) | 13; 15 number of MIH affected molars (As units: 6 MIH affected molars failures to attend follow up at 12 months which involved 6 participants) | 15; 16 number of MIH affected molars (As units: 5 MIH affected molars failures to attend follow up at 12 months which involved 5 participants)
Completed | 11; 13 number of MIH affected molars | 13; 15 number of MIH affected molars | 15; 16 number of MIH affected molars
Not Completed | 7; 8 number of MIH affected molars | 6; 6 number of MIH affected molars | 5; 5 number of MIH affected molars
Not completed — Lost to Follow-up | 7 | 6 | 5

BASELINE CHARACTERISTICS:
Population: MIH affected molars represent the number of participants analysed for each treatment interventions.This is because one participant can have more than one MIH affected molars assigned into the same or different treatment groups. The total number of participants involved in this study was 38 with 63 MIH affected molars involved. Total number of participants at baseline (1 participants may have >1 MIH molars into same or different group) assigned into all interventions was 57.
Units Other Than Participants: MIH affected molars
Groups:
- High Viscosity GIC (HVGIC): High Viscosity GIC
  High Viscosity Glass Ionomer Cement: The molar will be restored with HVGIC
- Silver Diamine Fluoride (SDF) + HVGIC: SDF and High Viscosity GIC
  Silver Diamine Fluoride: A single application of SDF 38% (Riva Star) on dry affected molar for 1 minute and immediately restored using HVGIC
- Papain Based Gel + SDF + HVGIC: SDF, Papain-Based Gel and High Viscosity GIC
  Papain-Based Gel: Papain based Gel (Papacare Duo) will be applied to the MIH affected molar for 60 seconds and repeated if required. The molar will be treated with SDF and restored using HVGIC
- Total: Total of all reporting groups
Arm/Group | High Viscosity GIC (HVGIC) | Silver Diamine Fluoride (SDF) + HVGIC | Papain Based Gel + SDF + HVGIC | Total
Number analyzed (Participants) | 18 | 19 | 20 | 57
Number analyzed (MIH affected molars) | 21 | 21 | 21 | 63
Age, Customized [Mean (Standard Deviation); unit: years] | 10.1 (2.80) | 7.9 (1.50) | 9.2 (2.44) | 9.2 (2.43)
Sex/Gender, Customized [Number; unit: participants]
  Male | 9 | 9 | 10 | 28
  Female | 12 | 12 | 11 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 18 | 19 | 20 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
MIH affected molars [Count of Participants; unit: Participants] — MIH affected molars were used to represent as baseline participants assigned into intervention group. 1 participants may have more than 1 MIH affected molars being assigned into the same or different intervention group.
  Participants | 18 | 19 | 20 | 57

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome Based on Success After Intervention on MIH Affected Molar at 6 Months
Description: Treated MIH affected molars must fulfilled all criteria for success in order to be reported as success. Criteria of 'Successful' on treated MIH affected molars include
  1. Absence of pain related to the treated tooth/teeth
  2. Absence of tenderness to percussion (TTP)
  3. No evidence of swelling of supporting soft tissue or presence of a sinus tract
  4. Absence of enamel breakdown and caries along margin of restoration
  5. Scale 0 and 1 for Schiff Cold Air Sensitivity Scale
Time Frame: 6 month
Population: Descriptive analysis of frequency was used. MIH affected molars represents as participants. This is because one participants may have more than 1 tooth assigned into one or more intervention groups.
Measure: Number; unit: number of Successful MIH affected molars
Units Other Than Participants: MIH affected molars
Arm/Group | High Viscosity GIC (HVGIC) | Silver Diamine Fluoride (SDF) + HVGIC | Papain Based Gel + SDF + HVGIC
Number analyzed (Participants) | 15 | 16 | 16
Number analyzed (MIH affected molars) | 18 | 18 | 17
number of Successful MIH affected molars | 17 | 18 | 17

2. Primary Outcome: Clinical Outcome Based on Success After Intervention on MIH Affected Molar at 12 Months
Description: Treated MIH affected molars must fulfilled all criteria for success in order to be reported as successful. Criteria of 'Successful' on treated MIH affected molars include
  1. Absence of pain related to the treated tooth/teeth
  2. Absence of tenderness to percussion (TTP)
  3. No evidence of swelling of supporting soft tissue or presence of a sinus tract
  4. Absence of enamel breakdown and caries along margin of restoration
  5. Scale 0 and 1 for Schiff Cold Air Sensitivity Scale
Time Frame: 12 month
Population: Descriptive analysis of frequency was used. MIH affected molars represent as participants in this analysis. This is because one participants may have more than 1 tooth assigned into one or more intervention groups.
Measure: Number; unit: number of successful MIH affected molars
Units Other Than Participants: MIH affected molars
Groups:
- Silver Diamine Fluoride (SDF ) + HVGIC: Silver Diamine Fluoride: A single application of SDF 38% (Riva Star) on dry affected molar for 1 minute and immediately restored using HVGIC
Arm/Group | High Viscosity GIC (HVGIC) | Silver Diamine Fluoride (SDF ) + HVGIC | Papain Based Gel + SDF + HVGIC
Number analyzed (Participants) | 12 | 11 | 14
Number analyzed (MIH affected molars) | 14 | 13 | 15
number of successful MIH affected molars | 14 | 13 | 15
Statistical Analysis 1: Comparison: High Viscosity GIC (HVGIC) vs Silver Diamine Fluoride (SDF ) + HVGIC vs Papain Based Gel + SDF + HVGIC; Test type: Other; p < 0.05, t-test, 2 sided; Odds Ratio (OR) = 0.7
Statistical Analysis 2: Comparison: High Viscosity GIC (HVGIC) vs Silver Diamine Fluoride (SDF ) + HVGIC vs Papain Based Gel + SDF + HVGIC; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: through study completion with an average of 1 year.
Groups:
- High Viscosity Glass Ionomer Cement (HVGIC): High Viscosity Glass Ionomer Cement (HVGIC): The MIH affected molar will be restored with HVGIC
Arm/Group | High Viscosity Glass Ionomer Cement (HVGIC) | Silver Diamine Fluoride (SDF) + HVGIC | Papain Based Gel + SDF + HVGIC
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/20

LIMITATIONS AND CAVEATS:
Small sample size of participants had led the result of this study to be interpreted with caution by other researchers. Ideal randomisation process cannot be fulfilled and MIH affected molars has been used as a unit for analyses. Thus, one participant may be assigned to more than one intervention groups. This situation pose a challenge to researcher as if one participant lost to follow up it will affect the number of unit/data to be analysed for each intervention groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT04710927/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT04710927/ICF_000.pdf